CLINICAL TRIAL: NCT05340127
Title: Summative Usability Study of a Novel Device - CEREBO® for Non Invasive Detection of Intracranial Haemorrhage
Brief Title: Summative Usability Study of CEREBO® - a Non Invasive Intracranial Hemorrhage Detector
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bioscan Research Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BR/US/2022/001
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Usability
Keywords: Ease of Use; Ease of learning; Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects examined by the study participants using CEREBO® (Experimental): CEREBO® - A non-invasive intracranial haemorrhage detector
  Scan Duration - 40 seconds per subject
  Frequency - Every operator will perform CEREBO® scan on at least 10 different subjects
  Adverse Effect: None
  Interventions: Device: CEREBO®

INTERVENTIONS:
Device: CEREBO® — Usability Study

SUMMARY:
Traumatic brain injury is one of the most common reasons for visits to the Emergency Department. More than 90% of patients who have suffered from head trauma present with a mild traumatic brain injury. Most of these patients do not present any symptom at the time of diagnosis thus delaying the detection. CEREBO®, a non-invasive, portable, rapid, point-of-care intracranial haemorrhage detector can avoid delayed detection by decreasing the time from injury to the initial CT scan. The study aims at assessing the summative usability of the device by determining its ease of use, ease of learning and satisfaction among the medical health professionals. The participants will be trained before the study and will be assessed periodically. Each participant will use the device on at least 10 subjects.

DETAILED DESCRIPTION:
A prospective interventional study designed to assess the summative usability and rapidity of CEREBO® - a portable device to detect intracranial haemorrhage. 10 participants from a Primary Health Centre will be enrolled in this study. The participants will be trained by the study staff before the study. The participant will fill in a questionnaire periodically. At the end of the study, the statistical analysis will be performed on the recorded data to establish the ease of use, ease of learning and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Operators

* Medical health professionals >18 years of age with a valid medical license to practice medicine belonging to one of the following categories and have given a written consent to participate in the study.
* MBBS
* Ayush
* Nurse
* Others

Subjects

* Of all ages and gender, have understood the study and gave a written informed consent.

Exclusion Criteria:

Subjects

* Cognitively impaired subjects unable to understand the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-20 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
To assess the usability of CEREBO® to detect intracranial haemorrhage | 2 week
  A questionnaire filled by the participants will be assessed by the study team to assess the ease of use, ease of learning and satisfaction

SECONDARY OUTCOMES:
To assess the rapidity of CEREBO® to detect intracranial haemorrhage | 2 week
  The time to perform the CEREBO® scan per subject will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Kaushik Vitthlapara, Principal Investigator — PHC, India

IPD SHARING:
Plan to Share IPD: No